CLINICAL TRIAL: NCT04557202
Title: Effect of Perioperative Selective alpha1-blockers in Non-stented Ureteroscopic Laser Lithotripsy for Ureteric Stones
Brief Title: Effect of Perioperative Selective alpha1-blockers in Non-stented Ureteroscopic Laser Lithotripsy for Ureteric Stones: A Randomized Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Maher Gamil Ahmed Higazy, assistant lecturer of Urology - ain shams university, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: fwa00001989
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Non-stented Ureteroscopic Laser Lithotripsy for Ureteric Stones
Keywords: Uretroscopic lithotripsy; non-stented; alpha1-blocker; LUTS; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: We enrolled 120 patients with lower ureteric stones. They were randomly divided into two groups. Group A had 58 patients who underwent non-stented ureteroscopy using Ho-YAG laser for stone disintegration and received alpha1-blockers for one week preoperatively and another two weeks postoperatively, while Group B had 62 patients who underwent non-stented ureteroscopy and laser and received placebo.
Who Masked: Participant, Outcomes Assessor
Masking Description: patients were blinded to the type of intervention, as well as the data collector
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A had 58 patients who underwent non-stented ureteroscopy using Ho-YAG laser for stone disintegration and received alpha1-blockers for one week preoperatively and another two weeks postoperatively
  Interventions: Drug: Tamsulosin Oral Capsule
- Group B (Placebo Comparator): 62 patients who underwent non-stented ureteroscopy and laser and received placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamsulosin Oral Capsule — To assess the efficacy of peri-operative alpha1 blockers on improving the success rate and decreasing complications of non-stented ureteroscopic laser lithotripsy for ureteric stones.
  Arms: Group A
Drug: Placebo — Placebo - control group
  Arms: Group B

SUMMARY:
To assess the efficacy of peri-operative alpha1 blockers on improving the success rate and decreasing complications of non-stented ureteroscopic laser lithotripsy for ureteric stones.

DETAILED DESCRIPTION:
Objective: To assess the efficacy of peri-operative alpha1 blockers on improving the success rate and decreasing complications of non-stented ureteroscopic laser lithotripsy for ureteric stones.

Patients and Methods: A randomized control trial was conducted at two high volume urological centers from September 2017 to December 2018. We enrolled 120 patients with lower ureteric stones. They were randomly divided into two groups. Group A had 58 patients who underwent non-stented ureteroscopy using Ho-YAG laser for stone disintegration and received alpha1-blockers for one week preoperatively and another two weeks postoperatively, while Group B had 62 patients who underwent non-stented ureteroscopy and laser and received placebo.

ELIGIBILITY:
Inclusion Criteria:

* patients with single lower ureteric stones of size range between 0.5 and 2 cm

Exclusion Criteria:

* Patients under the age of 18, pregnant women, or those with urinary tract infections, uncorrected bleeding disorders or coagulopathies, bilateral ureteric stones, single kidney, ureteral stricture, multiple ipsilateral ureteric stones were excluded from our study. Also, any patients who required ureteric stenting were excluded from our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Need for dilatation | intraoperative assessment
  ( to evaluate whether the ureteroscope will pass easily through the ureter if not , serial ureteric dilatation will be done and documented ) it is a yes or no evaluation

SECONDARY OUTCOMES:
Time of operation (min) | intraoperative assessment
  duration of the procedure in minutes
Lower urinary tract symptoms "LUTs" | early postoperative period ( 2 weeks)
  (frequency, urgency and dysuria) (Yes/NO)
Need for analgesia | first day postoperative
  need for analgesics for postoperative pain according to the numeric rating scale (yes/no)
Gross Hematuria | first day postoperative
  post operative hematuria (present or not )
Fever | early postoperative (2 weeks)
  elevated body temperature post operative in degree Celsius
hospital stay | from few hours up to 2 days postoperative
  duration in hours

CONTACTS AND LOCATIONS:
Locations (1):
- Urology department - ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided